CLINICAL TRIAL: NCT03587051
Title: Endurance Training and Post-exercise Low Glycemic Index Recovery Diet for Improving Postprandial Triglycerides
Brief Title: Low Versus High-glycemic Index Post-exercise Diets for Improving Metabolism and Body Composition
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Saskatchewan (Other)
Collaborators: Heart and Stroke Foundation of Canada (Other)
Responsible Party: Principal Investigator, Phil Chilibeck, Professor, University of Saskatchewan
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 17-171
Record Dates: First submitted 2018-06-27; First posted 2018-07-16 (Actual); Last update posted 2020-06-11 (Actual); Status verified 2020-06

CONDITIONS: Hypercholesterolemia
MeSH Terms: conditions — Hypercholesterolemia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Low glycemic index post-exercise diet (Experimental): Lentil-based post-exercise meal
  Interventions: Dietary Supplement: Low glycemic index post-exercise diet
- High glycemic index post-exercise diet (Active Comparator): Instant potato, white bread, and egg white post-exercise meal
  Interventions: Dietary Supplement: High glycemic index post-exercise diet

INTERVENTIONS:
Dietary Supplement: Low glycemic index post-exercise diet — Feeding of a low-glycemic index, lentil meal after 90 minutes of walking exercise
  Arms: Low glycemic index post-exercise diet
Dietary Supplement: High glycemic index post-exercise diet — Feeding of a high-glycemic index meal (i.e. instant mashed potatoes, white bread, egg whites) after 90 minutes of walking exercise
  Arms: High glycemic index post-exercise diet

SUMMARY:
Postprandial triglycerides are a strong risk factor for heart disease. The purpose is to assess the effects of a low-glycemic versus high-glycemic meal after 90 minute exercise sessions that are done 4 times a week for 6 weeks on postprandial triglyceride level. Secondary measurements include other lipids and body composition.

DETAILED DESCRIPTION:
The increase in triglycerides after a meal (i.e. postprandial triglycerides) is a strong risk factor for cardiovascular disease. Overweight/obese individuals have a greater triglyceride response to the same meal compared to lean individuals; therefore they are at greater risk. If exercise is performed the evening before a high-fat breakfast, the postprandial levels of triglycerides after the breakfast are reduced; however, if high glycemic index (GI) foods are consumed after the exercise session, the benefits of exercise on next-day postprandial triglycerides is negated. The investigators recently showed (HSFC funded) that consuming low GI foods after exercise is similar to fasting after exercise and superior to consumption of high GI foods for lowering next-day postprandial triglycerides. Low GI food was also superior for increasing fat oxidation, and lowering insulin, and low and very low density lipoproteins and preventing a decrease in high density lipoproteins. The benefits of an acute exercise session followed by low GI food consumption is now clear; however, it is not known whether this practice over weeks of exercise training results in accumulated and sustained benefits.

The purpose of this study is to determine the chronic effects of consuming low compared to high GI foods after exercise sessions over six weeks in overweight and obese individuals.

Twenty-four overweight and obese males and females will be randomized to consume either high or low GI foods immediately after exercise sessions (four sessions per week, 90 minutes per session, six weeks). At all other times of the day over the six weeks, they will be supplied a moderate GI diet, with calories and macronutrients based on four-day food diaries completed before the study. Two weeks before the intervention, participants will be required to go on the moderate GI diet, as a lead-in. One week into the lead-in, a baseline test will be done to determine postprandial metabolic responses (i.e. triglycerides, low and very low density lipoproteins, high density lipoproteins, insulin, and fat oxidation) after a morning high-fat breakfast. A week later, the same postprandial testing will be carried out the morning after the first exercise and post-exercise consumption of a low or high GI recovery meal. Participants will continue the training and post-exercise food consumption for the next six weeks, with postprandial measures taken again following the final exercise and feeding session. Body composition and aerobic fitness will be determined before and after the six week intervention.

The investigators hypothesize that the low GI post-exercise feeding will be superior to the high GI post-exercise feeding for reducing body fat, improving fat oxidation, and reducing postprandial triglycerides, insulin and other harmful lipids. The results of the study will provide clinicians, exercise professionals and dietitians unique and experimentally tested strategies for their clients to lose body fat and improve metabolic profiles, to reduce the risk of heart disease.

ELIGIBILITY:
Inclusion Criteria:

* Overweight or obese (BMI 25 or greater)

Exclusion Criteria:

* Smokers
* Diabetic
* Taking medications that affect carbohydrate or lipid metabolism

Ages: 18 Years to 44 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 25 (Actual)
Dates: Start 2018-07-15 (Actual); Primary Completion 2019-09-30 (Actual); Study Completion 2019-12-30 (Actual)

PRIMARY OUTCOMES:
Postprandial triglycerides | Change from baseline to 1 week and 6 weeks
  Triglyceride from serum

SECONDARY OUTCOMES:
Postprandial cholesterol | Change from baseline to 1 week and 6 weeks
  Cholesterol from serum
Postprandial low density lipoprotein | Change from baseline to 1 week and 6 weeks
  Low density lipoprotein from serum
Postprandial high density lipoprotein | Change from baseline to 1 week and 6 weeks
  High density lipoprotein from serum
Postprandial glucose | Change from baseline to 1 week and 6 weeks
  Glucose from serum
Postprandial insulin | Change from baseline to 1 week and 6 weeks
  Insulin from serum
Fasting Triglyceride | Change from baseline to 1 week and 6 weeks
  Triglyceride from serum
Fasting cholesterol | Change from baseline to 1 week and 6 weeks
  Cholesterol from serum
Fasting LDL-cholesterol | Change from baseline to 1 week and 6 weeks
  LDL from serum
Fasting HDL-cholesterol | Change from baseline to 1 week and 6 weeks
  HDL from serum
Fasting glucose | Change from baseline to 1 week and 6 weeks
  Glucose from serum
Fasting Insulin | Change from baseline to 1 week and 6 weeks
  Insulin from serum
Postprandial fat oxidation | Change from baseline to 1 week and 6 weeks
  Fat oxidation assessed by expiratory gases
Fat mass | Change from baseline to 6 weeks
  Fat mass assessed by dual energy x-ray absorptiometry
Waist Girth | Change from baseline to 6 weeks
  Waist girth assessed by a measurement tape

CONTACTS AND LOCATIONS:
Locations (1):
- University of Saskatchewan, Saskatoon, Saskatchewan, Canada

IPD SHARING:
Plan to Share IPD: No